CLINICAL TRIAL: NCT03358277
Title: Aripiprazole Added on Methylphenidate in the Treatment of Youths With Comorbid ADHD and DMDD
Brief Title: Aripiprazole Added on for DMDD in Youths With ADHD
Acronym: AAOFDIYWA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chin-Bin Yeh, MD, PhD, Director of Department of Psychiatry, Tri-Service General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSGH 099-05-159
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Disruptive Mood Dysregulation Disorder
MeSH Terms: interventions — 5,10-dihydro-5-methylphenazine; Methylphenidate; Aripiprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADHD+DMDD Group (Experimental): The subjects with comorbid ADHD and DMDD received pharmacological intervention with combination treatment of MPH+ APZ with flexible dosage according to clinical judgment for six weeks.
  Interventions: Drug: MPH + APZ

INTERVENTIONS:
Drug: MPH + APZ — MPH was administered with either Ritalin (from 10mg/day to 40mg/day) or Concerta (from 18mg/day to 36mg/day) according to clinical judgement for six weeks. APZ was administered with dose from 2.5mg/day to 5mg/day according to clinical judgement for six weeks.
  Other Names: MPH (Ritalin, Concerta), APZ (Abilify)

SUMMARY:
Objectives:

1. To investigate the effectiveness of adjuvant with aripiprazole to methylphenidate for disruptive mood dysregulation disorder (DMDD) in youths with attention-deficit/hyperactivity disorder (ADHD)
2. To investigate the neural basis of chronic irritability in youths with functional magnetic resonance imaging (fMRI)
3. To compare the clinical characteristics of youths with comorbid ADHD and DMDD to youths with ADHD only

DETAILED DESCRIPTION:
Background:

Disruptive mood dysregulation disorder (DMDD) in children and adolescents with attention-deficit/hyperactivity disorder (ADHD) is a common clinical challenge and leads to severe impact and burden on both the patients and their family. Although methylphenidate (MPH) showed good efficacy in the treatment of ADHD, there is still lack of well-established pharmacological treatment for DMDD. Furthermore, little research focuses on the effect of pharmacological treatment on neural correlates of chronic irritability. Previous literature suggested the potential role of atypical antipsychotics in the treatment of DMDD. Therefore, this study aimed to investigate the effectiveness of adjuvant of aripiprazole (APZ) to MPH in patients with comorbid ADHD and DMDD. In addition, the investigators explored the clinical manifestation and neural basis of DMDD using inventories, neuropsychological tests and neuroimaging studies.

Methods:

The investigators enrolled patients with ADHD+DMDD (n = 31) and ADHD only (n = 27). Those subjects were evaluated with inventories of emotional and behavioral problems, neuropsychological tests, as well as fMRI with challenging tests which aimed to induce frustration at baseline assessment. Then, subjects of ADHD+DMDD group received 6 weeks' combination treatment of MPH+ APZ with flexible dosage according to clinical judgment. All the initial evaluations were administered again after treatment. The comparison of clinical characteristics and neuroimaging findings between ADHD+DMDD group and ADHD only group will be conducted. In addition, the effectiveness of treatment will be analyzed. The effects of pharmacological treatment on neural correlates of chronic irritability will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

For subjects with comorbid ADHD and DMDD:

* Subject meets the DSM-5 criteria for ADHD and DMDD
* Subject is free from prior psychotropic medication for at least one year

For subjects with ADHD only :

* Subject meets the DSM-5 criteria for ADHD and DMDD
* Subject is free from prior psychotropic medication for at least one year

Exclusion Criteria:

* Patients not willing to participate in the study after detailed explanation
* Patients who could not follow the investigator's instructions
* Patients with severe neurological or mental illness such as epileptic disorder, schizophrenia, bipolar disorder, mental retardation or uncontrolled suicide risk
* Patients with severe medical illness or surgical conditions which were judged by investigators for safety concerns as inappropriate for this study, such as uncontrolled abnormal thyroid function, history of heart attack, uncontrolled hypertension.
* Patients taking psychotropic medication within one year prior to the evaluation for entering our study
* Patients being allergic to methylphenidate or aripiprazole
* Female patients being pregnant, nursing, or lactating

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-08-12 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist (CBCL) subscale scores | six weeks
  The Child Behavior Checklist (CBCL) is a widely used caregiver report form identifying problem behavior in children. The patient is rated on 113 items scored on a 3-point Likert-type scale. CBCL consists of eight empirically-based syndrome subscales. The range of subscale scores (summed) are: Aggressive Behavior (0-36), Anxious/Depressed (0-26), Attention Problems (0-20), Rule-Breaking Behavior (0-34), Somatic Complaints (0-22), Social Problems (0-22), Thought Problems (0-30), and Withdrawn/Depressed (0-16). The higher score suggests the more severe symptoms.

SECONDARY OUTCOMES:
Swanson, Nolan, and Pelham Scale-version IV (SNAP-IV) total and subscale scores | six weeks
  The SNAP-IV is a widely used caregiver report form identifying Attention-Deficit/Hyperactivity Disorder (ADHD) symptoms in children. The patient is rated on 26 items scored on a 4-point Likert-type scale. SNAP-IV consists of three subscales: inattention (items #1-#9, range of subscale summed score 0-27), hyperactivity/ impulsivity (items #11-#18, range of subscale summed score 0-27), and symptoms of Oppositional Defiant Disorder (items #19-#26, range of subscale summed score 0-24). The higher score suggests the more severe symptoms.
Beck Youth Inventories-II subscale scores | six weeks
  An self-reported inventory to evaluate children's and adolescents' emotional and social impairment. It includes five subscales: depression, anxiety, anger, disruptive behaviour, and self-concept. Each subscale consists of 20 items, and each item is scored on a 4-point Likert-type scale. The range of each subscale scores (summed) is 0-60. The higher score suggests the more severe symptoms.
Conner's Continuous Performance Test | six weeks
  A task-based computerized assessment of attention problems and neurological functioning
Children Color Trail Test (CCTT) | six weeks
  The CCTT assesses sustained attention, sequencing, and other executive functions.
Resting state functional magnetic resonance imaging | six weeks
  A method of functional brain imaging that can be used to evaluate regional interactions that occur when a subject is not performing an explicit task.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Bin Yeh, MD, PhD, Principal Investigator — Tri-Service General Hospital, National Defense Medical Center

IPD SHARING:
Plan to Share IPD: No